CLINICAL TRIAL: NCT01406691
Title: Treating Sleep Disruption in Teens With Millisecond Light Exposure During Sleep
Brief Title: Light Flashes to Treat Delayed Sleep Phase Disorder (DSPD)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Professor, Stanford University
Organization: VA Palo Alto Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kidflash; R01HD102344-01A1 (NIH)
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Delayed Sleep Phase Disorder
Keywords: sleep; delayed sleep phase disorder; circadian; teen; adolescent

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Light (Experimental): one hour of a sequence of light flashes (4000 lux, 3 msec, every 30 seconds); occurs during hour immediately prior to desired waketime
  Interventions: Device: Flashes
- Fake light (Placebo Comparator): during hour immediately prior to desired waketime, subjects will receive one light flash (insufficient to cause phase shift)
  Interventions: Device: Flashes

INTERVENTIONS:
Device: Flashes — one hour of a sequence of light flashes (4000 lux, 3 msec, every 30 seconds); occurs during the hour immediately prior to desired waketime

SUMMARY:
Delayed Sleep Phase Disorder (DSPD) is a sleep disruption that commonly occurs in teens and manifests as a difficulty in waking up in the morning, going to sleep early enough at night, and daytime disturbances such as depression, fatigue, and restlessness. The purpose of this study is to determine if brief flashes of light, that are scheduled to occur during sleep, are effective in treating DSPD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Full-time in high school
* primary sleep complaint consistent with delayed sleep phase disorder

Exclusion Criteria:

* sleep only in prone position
* currently taking medications specifically for the treatment of a sleep disorder

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | weekly for four weeks
  Determined by questionnaire (Adolescent Sleep Wake Scale)

SECONDARY OUTCOMES:
Mood | at the begining and end of intervention (4 weeks)
  Center for Epidemiologic Studies Depression Scale for Children (depressive symptoms) SNAP-IV 26 (ADHD symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Background] Zeitzer JM, Ruby NF, Fisicaro RA, Heller HC. Response of the human circadian system to millisecond flashes of light. PLoS One. 2011;6(7):e22078. doi: 10.1371/journal.pone.0022078. Epub 2011 Jul 8. PMID 21760955
- [Background] Zeitzer JM, Fisicaro RA, Ruby NF, Heller HC. Millisecond flashes of light phase delay the human circadian clock during sleep. J Biol Rhythms. 2014 Oct;29(5):370-6. doi: 10.1177/0748730414546532. Epub 2014 Sep 16. PMID 25227334
- [Background] Joyce DS, Spitschan M, Zeitzer JM. Optimizing Light Flash Sequence Duration to Shift Human Circadian Phase. Biology (Basel). 2022 Dec 13;11(12):1807. doi: 10.3390/biology11121807. PMID 36552316
- [Background] Joyce DS, Spitschan M, Zeitzer JM. Duration invariance and intensity dependence of the human circadian system phase shifting response to brief light flashes. Proc Biol Sci. 2022 Mar 9;289(1970):20211943. doi: 10.1098/rspb.2021.1943. Epub 2022 Mar 9. PMID 35259981
- [Result] Kaplan KA, Mashash M, Williams R, Batchelder H, Starr-Glass L, Zeitzer JM. Effect of Light Flashes vs Sham Therapy During Sleep With Adjunct Cognitive Behavioral Therapy on Sleep Quality Among Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e1911944. doi: 10.1001/jamanetworkopen.2019.11944. PMID 31553469